CLINICAL TRIAL: NCT00409461
Title: Comparison of Sirolimus Alone With Sirolimus Plus Tacrolimus in Type 1 Diabetic Recipients of Cultured Islet Cell Grafts
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: AZ-VUB (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other); Belgian Government (Other Government)
Allocation: Non-Randomized | Model: Factorial | Masking: None
Other Study IDs: 4-2001-434; G.0375.00; G.0084.02; GOA/2004/10
Record Dates: First submitted 2006-12-08; First posted 2006-12-11 (Estimated); Last update posted 2006-12-11 (Estimated); Status verified 2006-12

CONDITIONS: Islet Transplantation; Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

INTERVENTIONS:
Drug: ATG-Sirolimus-Tacrolimus

SUMMARY:
Proof of concept study in islet transplantation, two treatment arms (ATG SIR-TAC versus ATG SIR) each consisting of ten type 1 diabetic patients

ELIGIBILITY:
Inclusion Criteria:

* Type 1 insulin-dependent diabetic patients
* C-peptide < 0.15 nmol/l (<0.45 µg/l) 6 min. after glucagon IV (1mg) (glycemia > 180 mg/dl)
* diabetic nephropathy
* hypoglycaemic unawareness

Exclusion Criteria:

* smoker before transplantation
* plasma creatinine > 2 mg/dl
* albuminuria >1000 mg/24 hrs
* abnormal liver function
* history of thrombosis or pulmonary embolism
* history of malignancy, tuberculosis or chronic viral hepatitis
* history of any other serious illness which could be relevant for the protocol
* HLA antibodies
* EBV antibody negative
* HIV 1 & 2 antibody positive

Ages: 18 Years to 65 Years
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Bart Keymeulen, MD, PhD, Principal Investigator — AZ-VUB
Locations (2):
- Belgium (2):
  - Academisch Ziekenhuis and Diabetes Research Center - Brussels Free University-VUB, Brussels
  - Department of Endocrinology and Nephrology, UZ Gasthuisberg, Katholieke Universiteit Leuven -KUL, Leuven

REFERENCES:
- [Derived] Gillard P, Ling Z, Mathieu C, Crenier L, Lannoo M, Maes B, Roep B, Gorus F, Pipeleers D, Keymeulen B. Comparison of sirolimus alone with sirolimus plus tacrolimus in type 1 diabetic recipients of cultured islet cell grafts. Transplantation. 2008 Jan 27;85(2):256-63. doi: 10.1097/TP.0b013e31815e8926. PMID 18212631